CLINICAL TRIAL: NCT02714283
Title: Comparative Effectiveness and Safety of Inhaled Corticosteroids and Antimicrobial Compounds for Non-CF Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Alabama at Birmingham (Other); National Jewish Health (Other); COPD Foundation (Other)
Responsible Party: Principal Investigator, Kevin Winthrop, Associate Professor, Divisions of Infectious Diseases, and Public Health and Preventive Medicine, Oregon Health and Science University
Other Study IDs: CER-1503-29191
Record Dates: First submitted 2016-03-15; First posted 2016-03-21 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Bronchiectasis
Keywords: nontuberculous mycobacteria; corticosteroids; macrolides; antibiotics
MeSH Terms: conditions — Bronchiectasis | interventions — Azithromycin; Erythromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-CF bronchiectasis patients: Complete national 2006-2014 Medicare data from Part A, B and D will be obtained from CMS. We will use bronchiectasis ICD-9 codes 494.0 and 494.1 to identify patients with bronchiectasis within Medicare. From this identified bronchiectasis cohort, we will exclude patients with cystic fibrosis (ICD-9 codes 277.00-277.09), HIV infection (042), and a history of organ transplant (V42.0, V42.1, V42.6, V42.7, V42.8).
  Interventions: Drug: inhaled corticosteroid therapy; Drug: macrolide therapy

INTERVENTIONS:
Drug: inhaled corticosteroid therapy — We will evaluate and compare the clinical effectiveness and safety of long-term inhaled corticosteroid and macrolide antimicrobial therapies
Drug: macrolide therapy — We will evaluate and compare the clinical effectiveness and safety of long-term inhaled corticosteroid and macrolide antimicrobial therapies
  Other Names: azithromycin; erythromycin

SUMMARY:
The purpose of this study is to provide patients and their physicians with greater understanding of the risks and benefits of commonly used therapies for treatment of non-CF bronchiectasis

DETAILED DESCRIPTION:
Non-CF bronchiectasis is a chronic inflammatory lung disease that is closely linked to pulmonary NTM disease. Both are rare but rising in incidence and disproportionately affect the elderly and women. Therapy of non-CF bronchiectasis aims to reduce inflammation via either ICS-induced immunosuppression or antibiotic-associated immunomodulation and/or suppression of pathogenic organisms. Both strategies, pursued long-term alone or some cases concomitantly, have inherent risks, and the relative risks and benefits of these differential approaches are poorly studied to date. Ultimately, our study will provide patients and their physicians with greater understanding of the risks and benefits of these therapeutic choices.

ELIGIBILITY:
Inclusion Criteria:

* Within Medicare data, indicated diagnosis of Bronchiectasis by a Pulmonologist (ICD-9 code 494.0 and/or 494.1)

Exclusion Criteria:

* cystic fibrosis diagnosis, HIV infection, history of organ transplant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients within Medicare with a diagnosis of bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 90089 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Winthrop, MD, MPH, Principal Investigator — Oregon Health and Science University; Emily Henkle, PhD, MPH, Study Director — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deyo RA, Cherkin DC, Ciol MA. Adapting a clinical comorbidity index for use with ICD-9-CM administrative databases. J Clin Epidemiol. 1992 Jun;45(6):613-9. doi: 10.1016/0895-4356(92)90133-8. PMID 1607900
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Henkle E, Curtis JR, Chen L, Chan B, Aksamit TR, Daley CL, Griffith DE, Winthrop KL. Comparative risks of chronic inhaled corticosteroids and macrolides for bronchiectasis. Eur Respir J. 2019 Jul 18;54(1):1801896. doi: 10.1183/13993003.01896-2018. Print 2019 Jul. PMID 31000676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Complete national 2006-2014 Medicare data from Part A, B and D (but not C) were obtained from Center for Medicare and Medicaid Services for patients with ICD-9-CM code 494.0 or 494.1 (bronchiectasis without or with acute exacerbation).
Pre-assignment Details: From the identified bronchiectasis cohort, we excluded patients with cystic fibrosis, HIV infection, or a history of organ transplant. Such patients are fundamentally different than non-CF bronchiectasis patients who lack these factors with regard to their risk for infection, hospitalization, and many of the outcomes under study in this proposal.
Groups:
- Inhaled Corticosteroids (ICS): New use was defined as the first prescription for a minimum 28 day ("chronic") supply of ICS after a clean period of 12 months with no chronic use of either exposure of interest. ICS included ICS alone or in combination with long-acting beta agonists.
- Macrolide Monotherapy: New use was defined as the first prescription for a minimum 28 day ("chronic") supply of macrolide monotherapy after a clean period of 12 months with no chronic use of either exposure of interest. Macrolide monotherapy was defined as oral azithromycin or erythromycin and no other chronic prescription within 30 days that could be associated with NTM therapy (ethambutol, a rifamycin, or a fluoroquinolone). Patients who did not start on macrolide monotherapy were excluded.
Period: Overall Study
Arm/Group | Inhaled Corticosteroids (ICS) | Macrolide Monotherapy
Started (Treatment episode start) | 83589 | 6500
Completed (Earliest date: death, 1st outcome occurrence, study end, lost coverage, treatment stop or switch) | 83589 | 6500
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Corticosteroids (ICS) | Macrolide Monotherapy | Total
Number analyzed (Participants) | 83589 | 6500 | 90089
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 83589 | 6500 | 90089
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56583 | 4750 | 61333
  Male | 27006 | 1750 | 28756
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 362 | 17 | 379
  Asian/Pacific Islander | 3353 | 160 | 3513
  Black or African-American | 5338 | 236 | 5574
  Hispanic | 5188 | 203 | 5391
  White (non-Hispanic) | 68508 | 5820 | 74328
  Other/Unknown | 840 | 64 | 904
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Midwest | 17129 | 1612 | 18741
  United States: Northeast | 18629 | 992 | 19621
  United States: South | 33289 | 2897 | 36186
  United States: West | 14542 | 999 | 15541
Residential category [Count of Participants; unit: Participants]
  Rural | 65261 | 4798 | 70059
  Metropolitan | 18328 | 1702 | 20030
Physician encounters in the 12 month prior to Baseline [Count of Participants; unit: Participants]
  0-7 | 24345 | 1482 | 25827
  8-12 | 20027 | 1526 | 21553
  13-19 | 20549 | 1771 | 22320
  20+ | 18668 | 1721 | 20389
Pulmonologist encounters in the prior 12 months before baseline [Count of Participants; unit: Participants]
  0 | 19013 | 692 | 19705
  1 | 15157 | 941 | 16098
  2 | 15437 | 1032 | 16469
  3 | 11025 | 1005 | 12030
  4 | 7232 | 724 | 7956
  5+ | 15725 | 2106 | 17831
Inpatient admissions in the 12 months prior to baseline [Count of Participants; unit: Participants]
  0 | 49795 | 4108 | 53903
  1 | 17943 | 1299 | 19242
  2+ | 15851 | 1093 | 16944
Hospitalized respiratory infections in the 12 months prior to baseline [Count of Participants; unit: Participants] | 9583 | 885 | 10468
Number of acute respiratory infections in the 12 months prior to baseline [Count of Participants; unit: Participants]
  0 | 40746 | 2478 | 43224
  1 | 20193 | 1384 | 21577
  2-3 | 15993 | 1499 | 17492
  4+ | 6657 | 1139 | 7796
Comorbidities (any history) [Count of Participants; unit: Participants]
  Allergic bronchopulmonary aspergillosis | 854 | 64 | 918
  Alpha-1 antitrypsin deficiency | 292 | 43 | 335
  Asthma | 33480 | 1795 | 35275
  COPD/emphysema | 70548 | 5050 | 75598
  Interstitial lung disease | 5526 | 507 | 6033
  Lung cancer | 3497 | 196 | 3693
  NTM History | 3164 | 1307 | 4471
  Primary ciliary dyskinesia | 141 | 23 | 164
  Primary immune deficiency | 3857 | 466 | 4323
  Pseudomonas infection | 5123 | 810 | 5933
  Silicosis | 103 | 6 | 109
Adapted Charlson comorbidity index (prior 12 months) [Count of Participants; unit: Participants] — Charlson comorbidity index, higher score is worse.
  Participants
    0 | 20514 | 1534 | 22048
    1 | 33959 | 3119 | 37078
    2+ | 29116 | 1847 | 30963

OUTCOME MEASURES:

1. Primary Outcome: Nontuberculous Mycobacterial (NTM) Disease
Description: Incidence of treated pulmonary nontuberculous mycobacterium (NTM) disease
Time Frame: up to 8 years
Population: Analysis population excluded all patients with a history of NTM treatment or diagnosis prior to exposure start.
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Inhaled Corticosteroids (ICS) | Macrolide Monotherapy
Number analyzed (Participants) | 16136 | 1496
Number analyzed (Patient-years) | 19460 | 1736
Events | 188 | 32
Statistical Analysis 1: Comparison: Inhaled Corticosteroids (ICS) vs Macrolide Monotherapy; Due to the small sample size in the macrolide monotherapy group, for this outcome, the results are considered exploratory/descriptive only; Test type: Superiority; p = 0.19, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.51 to 1.14] — ICS (numerator) compared to macrolide monotherapy (denominator)

2. Primary Outcome: Hospitalized Respiratory Infection
Description: Among a national cohort of non-CF bronchiectasis patients, we will compare the effectiveness of corticosteroid and macrolide therapy with regards to prevention of hospitalized respiratory infection.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Groups:
- Non-CF Bronchiectasis Patients on ICS Monotherapy: New use was defined as the first prescription for a minimum 28 day ("chronic") supply of ICS after a clean period of 12 months with no chronic use of either exposure of interest. ICS included ICS alone or in combination with long-acting beta agonists.
- Non-CF Bronchiectasis Patients on Macrolide Monotherapy: New use was defined as the first prescription for a minimum 28 day ("chronic") supply of macrolide monotherapy after a clean period of 12 months with no chronic use of either exposure of interest. Macrolide monotherapy was defined as oral azithromycin or erythromycin and no other chronic prescription within 30 days that could be associated with NTM therapy (ethambutol, a rifamycin, or a fluoroquinolone). Patients who did not start on macrolide monotherapy were excluded.
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 33328 | 3068
Events | 4213 | 317
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p < 0.0001, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.23 to 1.57] — ICS (numerator) compared to macrolide monotherapy (denominator)

3. Secondary Outcome: Sudden Cardiac Arrest
Description: Myocardial infarction event
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 34688 | 3171
Events | 892 | 81
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.21, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.67 to 1.09] — ICS (numerator) compared to macrolide monotherapy (denominator)

4. Secondary Outcome: Sensorineural Hearing Loss
Description: Sensorineural hearing loss.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Groups:
- Non-CF Bronchiectasis Patients on ICS Monotherapy: Patients prescribed a 28 day or more supply of ICS, with an absence of ICS prescriptions for at least the 12 months prior to identified prescription. ICS include beclomethasone, budesonide, flunisolide, fluticasone, mometasone, triamcinolone, ipratropium/albuterol, budesonide/formoterol, or fluticasone/salmeterol. Exclude baseline 28+ day macrolide, missing geographic or socioeconomic data.
- Non-CF Bronchiectasis Patients on Macrolide Monotherapy: Patients prescribed a 28 day or more supply of a macrolide, with an absence of macrolide prescriptions for at least the 12 months prior to identified prescription. Macrolides include oral azithromycin, clarithromycin, and erythromycin. Exclude baseline 28+ day ICS, missing geographic or socioeconomic data
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 33491 | 2993
Events | 2574 | 347
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p < 0.0001, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.64 to 0.82] — ICS (numerator) compared to macrolide monotherapy (denominator)

5. Secondary Outcome: Hip Fracture
Description: Hip fracture.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 34661 | 3173
Events | 919 | 77
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.87, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.80 to 1.32] — ICS (numerator) compared to macrolide monotherapy (denominator)

6. Secondary Outcome: Opportunistic Infections
Description: Opportunistic infections.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 34200 | 3113
Events | 1585 | 180
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.23, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.76 to 1.07] — ICS (numerator) compared to macrolide monotherapy (denominator)

7. Secondary Outcome: All-cause Mortality
Description: All-cause mortality.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 34912 | 3193
Events | 3362 | 270
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.20, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.96 to 1.25] — ICS (numerator) compared to macrolide monotherapy (denominator)

8. Secondary Outcome: All-cause Hospitalization
Description: All-cause hospitalization.
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 28882 | 2729
Events | 17939 | 1352
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p < 0.0001, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.08 to 1.21] — ICS (numerator) compared to macrolide monotherapy (denominator)

9. Secondary Outcome: Hemoptysis
Description: Hemoptysis event
Time Frame: up to 8 years
Measure: Number; unit: Events
Units Other Than Participants: Patient-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (Patient-years) | 34835 | 3185
Events | 253 | 31
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.99, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.66 to 1.51] — ICS (numerator) compared to macrolide monotherapy (denominator)

10. Secondary Outcome: Arrhythmia
Description: Arrhythmia (principal diagnosis)
Time Frame: up to 8 years
Measure: Number; unit: events
Units Other Than Participants: person-years
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
Number analyzed (Participants) | 83495 | 6498
Number analyzed (person-years) | 31395 | 2855
events | 9508 | 728
Statistical Analysis 1: Comparison: Non-CF Bronchiectasis Patients on ICS Monotherapy vs Non-CF Bronchiectasis Patients on Macrolide Monotherapy; Test type: Superiority; p = 0.0005, Regression, Cox; Adjusted for propensity score decile, oral corticosteroid use, and NTM history; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.07 to 1.25] — ICS (numerator) compared to macrolide monotherapy (denominator)

ADVERSE EVENTS:
Time Frame: This is a retrospective observational study. Only medical history data was collected.
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored. We report Safety Outcomes in the Outcomes section.
Arm/Group | Non-CF Bronchiectasis Patients on ICS Monotherapy | Non-CF Bronchiectasis Patients on Macrolide Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Claims-based data limits our ability to confirm bronchiectasis diagnoses and include disease symptoms/severity in our models. Results may not be applicable to <65 year old bronchiectasis patients who have a lower underlying risk of pneumonia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02714283/Prot_SAP_000.pdf